CLINICAL TRIAL: NCT05287230
Title: Developing a Trauma-focused Intervention for Older Adults Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Monique J. Brown, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00114522; K01MH115794 (NIH)
Record Dates: First submitted 2022-02-18; First posted 2022-03-18 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Trauma; Hiv; Aging
MeSH Terms: conditions — Wounds and Injuries; Acquired Immunodeficiency Syndrome | interventions — Coping Skills; Seroconversion; Aging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: CoSHA (Coping with childhood Sexual Abuse, HIV, and Aging)
- Control (Other)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: CoSHA (Coping with childhood Sexual Abuse, HIV, and Aging) — Investigators will use concepts from the LIFT and REFLECT interventions.
  Arms: Intervention
Behavioral: Control — Participants will watch HIV and health related videos and discuss how it is related to aging with HIV.
  Arms: Control

SUMMARY:
Investigators are adapting the LIFT and REFLECT interventions for older adults living with HIV who have been exposed to childhood sexual abuse.

ELIGIBILITY:
Inclusion Criteria:

* Living with HIV
* 50 years old or older
* <100 % ART adherence
* depressive symptoms

Exclusion Criteria:

* Not living with HIV
* <50 years
* 100% ART Adherence

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monique J Brown, PhD, MPH, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to other researchers.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available to other researchers after investigators have submitted the related primary paper.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 17 | 11
Completed | 13 | 6
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 17 | 11 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 11 | 28
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 17 | 10 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 6 | 20
  White | 2 | 4 | 6
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 11 | 28

OUTCOME MEASURES:

1. Primary Outcome: ART Adherence
Description: Investigators will measure number of participants who report improved adherence to antiretroviral therapy in the past month using the 30-day visual analogue scale (VAS). Minimum is 0, Maximum is 100%. Higher scores mean better ART adherence.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 17 | 11
score on a scale | 79.0 (25.9) | 92.7 (2.5)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other; p = 0.061, ANOVA — A priori threshold for statistical significance is p<0.05

2. Primary Outcome: ART Adherence
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 7
score on a scale | 92.4 (11.3) | 96.4 (4.8)

3. Primary Outcome: ART Adherence
Description: Investigators will measure number of participants who report improved adherence to antiretroviral therapy in the past month using the 30-day visual analogue scale (VAS)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 12 | 6
score on a scale | 79.1 (29.1) | 96.3 (4.3)

4. Primary Outcome: ART Adherence
Description: as for outcome 3
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 12 | 7
score on a scale | 83.7 (22.0) | 91.1 (22.6)

5. Secondary Outcome: Health-related Quality of Life - General Health
Description: Investigators will measure health-related quality of life of participants, specifically, general health, using the Centers for Disease Control and Prevention Health Days Core Module (CDC HRQOL-4). Minimum value is 1. Maximum value is 5. Values were recoded so that higher scores mean better outcome.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 17 | 11
score on a scale | 2.59 (0.80) | 2.36 (1.21)

6. Secondary Outcome: Health-related Quality of Life - General Health
Description: as for outcome 5
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 14 | 6
score on a scale | 2.64 (1.08) | 3.50 (1.05)

7. Secondary Outcome: Health-related Quality of Life - General Health
Description: as for outcome 5
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 13 | 7
score on a scale | 2.69 (0.75) | 3.29 (1.11)

8. Secondary Outcome: Health-related Quality of Life - General Health
Description: as for outcome 5
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 13 | 7
score on a scale | 2.85 (0.80) | 3.14 (1.21)

9. Other Pre Specified Outcome: Depressive Symptoms
Description: Investigators will measure depressive symptoms as measured by the Patient Health Questionnaire-9 which ranges from 0 to 24 with higher values representing greater depressive symptoms.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 16 | 11
score on a scale | 21.6 (7.7) | 22.8 (7.4)

10. Other Pre Specified Outcome: Depressive Symptoms
Description: as for outcome 9
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 14 | 7
score on a scale | 19.3 (7.7) | 18.0 (6.4)

11. Other Pre Specified Outcome: Depressive Symptoms
Description: as for outcome 9
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 13 | 7
score on a scale | 19.5 (8.7) | 18.6 (6.9)

12. Other Pre Specified Outcome: Depressive Symptoms
Description: as for outcome 9
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 13 | 7
score on a scale | 14.5 (5.0) | 18.1 (4.3)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Participants were not at risk for serious adverse events, mortality or other adverse events.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/11
Other Adverse Events (participants affected / at risk) | 0/17 | 0/11

LIMITATIONS AND CAVEATS:
Small sample size as this is a pilot trial. Therefore, results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT05287230/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT05287230/ICF_001.pdf